CLINICAL TRIAL: NCT06804239
Title: Improving Activity in Adults With Chronic Pain: Self-Directed Versus Guided Support With Online Resources
Brief Title: Improving Activity in Adults With Chronic Pain With Online Resources
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Marian Wilson, Associate Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20809
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Activity; Online resources
MeSH Terms: conditions — Chronic Pain; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a User Guide and weekly prompts with access to an Online Pain-Management Resource
  Interventions: Behavioral: User guide with prompts
- Active-control (Active Comparator): The active-control group receives access to the Online Pain-Management Resource, but no User Guide or prompts.
  Interventions: Behavioral: User guide with prompts

INTERVENTIONS:
Behavioral: User guide with prompts — A user guide and prompts to assist use of an Online Pain-Management Resource

SUMMARY:
A randomized controlled study will test whether adults with chronic pain have improved outcomes when receiving a User Guide and weekly prompts for a newly designed Online Pain-Management Resource when compared to an active-control group that receives access to the Online Pain-Management Resource, but no User Guide or prompts. Outcomes of interest include measures of activity, sleep, pain and level of use of the online pain-management resource.

DETAILED DESCRIPTION:
Participants with chronic pain will be randomized in this pilot study to an intervention group that receives a User Guide and weekly prompts to use an Online Pain-Management Resource or an active-control group that receives access to the Online Pain-Management Resource, but no User Guide or prompts. Outcomes of interest include:

i. Changes in activity and sleep over time when online resources are paired with using a wearable activity tracker (Fitbit Inspire 3®); ii. Self-reported pain and pain-related measures; and iii. Level of use of the online pain-management resource. All participants will also be asked to provide feedback on the online pain-management resource. The information collected throughout the study will inform the development team on the website's usefulness and whether guided use is superior to unguided self-directed use of the online pain resource.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* chronic pain at least 3 months
* interested in increasing activity level
* able to read and speak English
* reside within US
* willing to have activity tracker shipped to address
* able to download Fitbit app onto phone or computer
* willing to use Fitbit device for most days and nights during 8 weeks study

Exclusion Criteria:

* medical or psychological conditions that would prevent study participation
* planned surgery or procedure that would prevent study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Activity | 8 weeks
  Changes in activity as recorded on wearable activity tracker (Fitbit Inspire 3®)
Sleep | 8 weeks
  Changes in sleep as recorded on wearable activity tracker (Fitbit Inspire 3®)

SECONDARY OUTCOMES:
Pain intensity | 8 weeks
  Patient reported outcomes measurement information system (PROMIS) Pain Intensity measures 1a and 3A where higher value means worse pain (1-5 rating).
Pain Interference | 8 weeks
  Patient reported outcomes measurement information system (PROMIS) Pain Interference 8 item measure where higher value means worse pain (1-5 rating)
Chronic Pain Acceptance | 8 weeks
  Chronic Pain Acceptance Questionnaire is 14 items where 0=never true and 6=always true and higher scores indicate greater acceptance.
Kinesiophobia | 8 weeks
  Tampa Scale of Kinesiophobia 17 items measures fear of movement and pain where 1=strongly disagree and 4=strongly agree. Higher scores indicate greater fear of movement and pain. A score of 37 or higher is often considered indicative of clinically significant kinesiophobia.
Sleep disturbance | 8 weeks
  Patient reported outcome measurement information system (PROMIS) Sleep Disturbance Short Form 4a where 5= Very poor or not at all and 1= very good or very much. Higher scores indicate increased sleep disturbance.
System Usability | 8 weeks
  Pain hub system usability scale 10 items rating 1-5 about the ease of system use. Higher scores are more favorable usability ratings.
Client Satisfaction | 8 weeks
  Pain hub client satisfaction 8-item questionnaire rating items 1-4 where higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington State University College of Nursing, Spokane, Washington
  - Washington State University, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Interested persons can contact the PI for deidentified data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After study ends for 3 years
Access Criteria: People with a scientific rationale for requesting the information
URL: https://nursing.wsu.edu/directory/wsu-profile/marian.wilson/

REFERENCES:
- [Background] Ruehlman, L.S., Bindler, R.J., Rangel, T.L. et al. Perspectives of Adults with Pain Regarding Online Pain Self-Management Resources. J. technol. behav. sci. (2024). https://doi.org/10.1007/s41347-024-00433-7